CLINICAL TRIAL: NCT06764212
Title: Investigation of the Diagnostic Efficacy of the Amount of Fascial Sliding Measured by M-Mode Ultrasonography in the Diagnosis of Myofascial Pain Syndrome
Brief Title: Investigation of the Diagnostic Efficacy of the M-Mode Ultrasonography in the Diagnosis of Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BursaYIEAH-2019-6-24
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Myofascial Pain Syndromes
Keywords: pain; ultrasound
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mps (Active Comparator): M-mode ultrasonography images of the fascia under the trapezius muscle will be recorded during 3 different movements.
  Interventions: Diagnostic Test: Ultrasound
- healthy volunteers (Active Comparator): M-mode ultrasonography images of the fascia under the trapezius muscle will be recorded during 3 different movements.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — M-mode ultrasonography images of the fascia under the trapezius muscle will be recorded during 3 different movements.
  Other Names: M-Mode musculoskeletal ultrasound

SUMMARY:
Myofascial pain syndrome, or MPS, is a prevalent musculoskeletal disorder, which is characterised by the presence of muscle pain and tenderness. The inflammation and microtrauma that are the consequence result in adhesions between the fascial layers. It has been reported that these adhesions prevent the fasciae from sliding over each other and contribute to pain.

DETAILED DESCRIPTION:
The rhomboid and trapezius muscles are commonly involved in MPS, which often affects the upper extremity.

This study hypothesized that muscle sliding decreases in patients with MPS. To this end, the investigators measured the amount of fascial sliding of the trapezius muscle in healthy volunteers and patients with MPS using M-mode ultrasound and a software-assisted program to investigate the differences and diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

* At least one active trigger point
* Moderate back pain lasting more than 3 months
* Diagnosis of MPS according to Travell and Simons diagnostic criteria
* Healthy volunteers

Exclusion Criteria:

* cervical disc disease
* Fibromyalgia
* Central or peripheral nerve disease
* Shoulder joint disease
* Malignancy
* Rheumatic disease
* those who had been treated for MPS within 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
m-mode | 30 minutes
  The amount of displacement of the fascia under the Trapezius muscle during arm lift, neck lateral and anterior flexion, and shoulder lift in a sitting position and the M-mode ultrasonography image will be recorded. The measurements obtained from the recordings will be recorded.

SECONDARY OUTCOMES:
Trapezius and rhomboid muscle | 30 minutes
  Trapezius and rhomboid muscle thickness measurements will be made via ultrasound
vas | baseline
  Visual Analog Scale was used for pain. Pain intensity was measured using 0-10 cm visual analogue scale (VAS). The findings suggested that 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.
NPDS | baseline
  Neck and Disability Scale (NPDS):
  The 20-item Neck and Disability Scale is scored on a 10 cm visual analog scale and ranges from 0 to 5 points. The test aims to measure the impact of neck pain on quality of life, functionality, and disability
sf-12 | baseline
  The SF-12 form, which includes scales to assess physical (SF-12-PCS) and mental (SF-12-MCS) status, was created by taking 12 different items from 8 other titles of the SF-36, which is the extended version

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Burcu Metin Ökmen, Nilufer, Bursa
  - Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa